CLINICAL TRIAL: NCT05255653
Title: Refining Adjuvant Treatment in Endometrial Cancer Based on Molecular Features: the P53abn-RED Trial, the MMRd-GREEN Trial, the NSMP-ORANGE Trial and the POLEmut-BLUE Trial
Brief Title: Refining Adjuvant Treatment in Endometrial Cancer Based on Molecular Features
Acronym: RAINBO
Status: Recruiting | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: Leiden University Medical Center (Other)
Collaborators: Institute Gustave Roussy (sponsor p53abn-RED trial) (Unknown); Leiden University Medical center (sponsor MMRd-GREEN trial) (Unknown); University College London (sponsor NSMP-ORANGE trial) (Unknown); Canadian Clinical Trials Group (sponsor POLEmut-BLUE trial) (Unknown); Dutch Gynaecological Oncology Group (Other); Comprehensive Cancer Centre The Netherlands (Other); Cancer Research UK & UCL Cancer Trials Centre (Other); Dutch Cancer Society (Other); AstraZeneca (Industry); National Cancer Institute, France (Other Government); Canadian Institutes of Health Research (CIHR) (Other Government)
Responsible Party: Principal Investigator, Carien Creutzberg, prof, Leiden University Medical Center
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: RAINBO; ENGOT-en14-1,2,3,4 (Other: ENGOT); CCTG EN.10 TAPER arm A POLE (Other: CCTG (only for the POLEmut-BLUE trial))
Record Dates: First submitted 2022-02-01; First posted 2022-02-24 (Actual); Last update posted 2024-11-29 (Actual); Status verified 2024-10

CONDITIONS: Endometrial Cancer
Keywords: Endometrial Cancer; Molecular risk factors; Olaparib; Durvalumab; Progestagens; Chemoradiation; Radiotherapy; Observation; p53; MMRd; NSMP; POLE
MeSH Terms: conditions — Endometrial Neoplasms | interventions — olaparib; Drug Therapy; Cisplatin; Carboplatin; Paclitaxel; durvalumab; Medroxyprogesterone Acetate; Progestins; Megestrol Acetate; Observation

STUDY DESIGN:
Intervention Model Description: Platform trial wherein eligible patients are assigned to one of four parallel running clinical trials. Three of four trials are randomised controlled trials and one is a prospective clinical trial with two study arms.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (8):
- p53abn-RED trial: experimental (Experimental): Adjuvant radiotherapy and chemotherapy followed by olaparib (lynparza), 300 mg twice daily, for one year
  Interventions: Drug: Olaparib; Radiation: Pelvic external beam radiotherapy; Drug: Chemotherapy; Radiation: Vaginal brachytherapy
- p53abn-RED trial: control (Active Comparator): Adjuvant radiotherapy and chemotherapy
  Interventions: Radiation: Pelvic external beam radiotherapy; Drug: Chemotherapy; Radiation: Vaginal brachytherapy
- MMRd-GREEN trial: experimental (Experimental): Adjuvant radiotherapy combined with and followed by durvalumab, 1500 mg intravenous once every 4 weeks for in total 1 year (13 cycles)
  Interventions: Radiation: Pelvic external beam radiotherapy; Drug: Durvalumab; Radiation: Vaginal brachytherapy
- MMRd-GREEN trial: control (Active Comparator): Adjuvant pelvic external beam radiotherapy +/- chemotherapy
  Interventions: Radiation: Pelvic external beam radiotherapy; Drug: Chemotherapy; Radiation: Vaginal brachytherapy
- NSMP-ORANGE trial: experimental (Experimental): Adjuvant radiotherapy followed by oral progestagens (medroxyprogesterone acetate or megestrol acetate) for two years
  Interventions: Radiation: Pelvic external beam radiotherapy; Drug: Medroxyprogesterone Acetate; Drug: Megestrol Acetate; Radiation: Vaginal brachytherapy
- NSMP-ORANGE trial: control (Active Comparator): Adjuvant radiotherapy and chemotherapy
  Interventions: Radiation: Pelvic external beam radiotherapy; Drug: Chemotherapy; Radiation: Vaginal brachytherapy
- POLEmut-BLUE trial: main cohort (Other): No adjuvant therapy in women with:
  * stage IA (not confined to polyp), grade 3, pN0, with or without LVSI
  * stage IB, grade 1 or 2, pNx/N0, with or without LVSI
  * stage IB, grade 3, pN0, without substantial LVSI
  * stage II (microscopic), grade 1 or 2, pN0, without substantial LVSI
  Interventions: Other: Observation
- POLEmut-BLUE trial: exploratory cohort (Other): No adjuvant therapy or vaginal brachytherapy or pelvic external beam radiotherapy in women with:
  * stage IA grade 3 - stage III not included in main cohort of the POLEmut-BLUE trial
  * Multiple molecular classifiers Stage IA (not confined to polyp), grade 3 - Stage III
  Interventions: Radiation: Pelvic external beam radiotherapy; Radiation: Vaginal brachytherapy; Other: Observation

INTERVENTIONS:
Drug: Olaparib — 300 mg twice daily for one year
  Other Names: Lynparza
  Arms: p53abn-RED trial: experimental
Radiation: Pelvic external beam radiotherapy — 45.0-48.6 Gy; 1.8-2.0 Gy per fraction, 5 fractions a week
  Other Names: EBRT
  Arms: MMRd-GREEN trial: control; MMRd-GREEN trial: experimental; NSMP-ORANGE trial: control; NSMP-ORANGE trial: experimental; POLEmut-BLUE trial: exploratory cohort; p53abn-RED trial: control; p53abn-RED trial: experimental
Drug: Chemotherapy — Preferably concurrent and adjuvant according to the PORTEC-3 schedule: two cycles of intravenous cisplatin 50mg/m² in the first and fourth week of the pelvic external beam radiotherapy followed by four cycles of intravenous carboplatin AUC 5 and paclitaxel 175 mg/m² at 21-day intervals.
  Other Names: Cisplatin; Carboplatin; Paclitaxel
  Arms: MMRd-GREEN trial: control; NSMP-ORANGE trial: control; p53abn-RED trial: control; p53abn-RED trial: experimental
Drug: Durvalumab — 1500 mg intravenous once every 4 weeks for in total 1 year (13 cycles) starting within the first week of radiotherapy,
  Other Names: Imfinzi
  Arms: MMRd-GREEN trial: experimental
Drug: Medroxyprogesterone Acetate — Oral medroxyprogesterone acetate for two years
  Other Names: Progestogen
  Arms: NSMP-ORANGE trial: experimental
Drug: Megestrol Acetate — Oral medroxyprogesterone acetate for two years
  Other Names: Progestogen
  Arms: NSMP-ORANGE trial: experimental
Radiation: Vaginal brachytherapy — Vaginal brachytherapy is to be considered in patients with documented cervical stromal involvement and/or substantial LVSI. Brachytherapy is given with a vaginal cylinder or vaginal ovoids or ring applicator, according to the center's standard technique. When using a cylinder, the active length will ideally be 2-3 cm, with the reference isodose covering the proximal 2.5-3 cm of the vagina. High-dose-rate (HDR) and pulse-dose-rate (PDR) schedules are permitted, which deliver an EQD2 equivalent dose of 10-14 Gy at 5 mm from the vaginal mucosa (to obtain a cumulative EDQ2 of 60 Gy at 5 mm).
  Arms: MMRd-GREEN trial: control; MMRd-GREEN trial: experimental; NSMP-ORANGE trial: control; NSMP-ORANGE trial: experimental; POLEmut-BLUE trial: exploratory cohort; p53abn-RED trial: control; p53abn-RED trial: experimental
Other: Observation — No adjuvant therapy
  Arms: POLEmut-BLUE trial: exploratory cohort; POLEmut-BLUE trial: main cohort

SUMMARY:
The RAINBO umbrella program consists of four clinical trials investigating new adjuvant therapies in endometrial cancer patients. Eligible patients will be assigned to one of the four RAINBO trials based on the molecular profile of their cancer:

* p53 abnormal endometrial cancer patients to the p53abn-RED trial
* mismatch repair deficient endometrial cancer patients to the MMRd-GREEN trial
* no specific molecular profile endometrial cancer patients to NSMP-ORANGE trial
* POLE mutant endometrial cancer patients to the POLEmut-BLUE trial

DETAILED DESCRIPTION:
The p53abn-RED trial (NCT05255653-1) is an international, multicenter, phase III randomised trial wherein adjuvant chemoradiation followed by olaparib for one year is compared to adjuvant chemoradiation.

The MMRd-GREEN trial (NCT05255653-2) is an international, multicenter, phase III randomised trial wherein adjuvant pelvic external beam radiotherapy combined with and followed by durvalumab for one year is compared to adjuvant pelvic external beam radiotherapy with or without chemotherapy.

The NSMP-ORANGE trial (NCT05255653-3) is an international, multicenter, phase III randomised trial wherein adjuvant pelvic external beam radiotherapy followed by progestogens for two years is compared to adjuvant chemoradiation.

The POLEmut-BLUE trial (NCT05255653-4) is an international, multicenter, single arm, phase II trial wherein safety of de-escalation of adjuvant therapy is investigated: no adjuvant therapy for stage I-II disease and no adjuvant therapy or pelvic external beam radiotherapy only for stage III disease.

The overarching RAINBO research project will combine the data and tumor material of the four RAINBO clinical trials to perform translational research and compare molecular profile-based adjuvant therapy to standard adjuvant therapy in terms of effectiveness, toxicity, quality of life and cost utility.

ELIGIBILITY:
Participants of the four RAINBO trials should be eligible according to the inclusion and exclusion criteria of both the overarching RAINBO trials program and the clinical trial that they are assigned to based on the molecular profile.

Inclusion Criteria of the overarching RAINBO program:

* Histologically confirmed diagnosis of endometrial cancer (EC) of the following histotypes: endometrioid endometrial carcinoma, serous endometrial carcinoma, uterine clear cell carcinoma, dedifferentiated and undifferentiated endometrial carcinoma, uterine carcinosarcoma and mixed endometrial carcinomas of the aforementioned histotypes.
* Full molecular classification performed following the diagnostic algorithm described in WHO 2020 (5th Edition, IARC, Lyon, 2020)
* Hysterectomy and bilateral salpingo-oophorectomy with or without lymphadenectomy or sentinel node biopsy, without macroscopic residual disease after surgery
* No distant metastases as determined by pre-surgical or post-surgical imaging (CT scan of chest, abdomen and pelvis or whole-body PET-CT scan)
* WHO performance status 0, 1 or 2
* Expected start of adjuvant treatment (if applicable) within 10 weeks after surgery
* Patients must be accessible for treatment and follow-up
* Written informed consent for participation in one of the RAINBO trials, permission for the contribution of a tissue block for translation research and permission for the use and sharing of data for the overarching research project according to the local Ethics Committee requirements.

Exclusion Criteria overarching RAINBO program:

* History of another primary malignancy, except for non-melanoma skin cancer, in the past 5 years
* Prior pelvic radiation

The p53abn-RED trial

Inclusion criteria:

* p53 abnormal EC
* Histologically confirmed stage I (with invasion) II or III EC
* WHO Performance score 0-1
* Body weight > 30 kg
* Adequate systemic organ function:

  * Creatinine clearance (> 40 cc/min): Measured creatinine clearance (CL) >40 mL/min or Calculated creatinine CL>40 mL/min by the Cockcroft-Gault formula (Cockcroft and Gault 1976) or by 24-hour urine collection for determination of creatinine clearance.
  * Adequate bone marrow function : hemoglobin >9.0 g/dl, Absolute neutrophil count (ANC) ≥1.0 x 109/l, platelet count ≥75 x 109/l.
  * Adequate liver function: bilirubin ≤1.5 x institutional upper limit of normal (ULN). This will not apply to patients with confirmed Gilbert's syndrome (persistent or recurrent hyperbilirubinemia that is predominantly unconjugated in the absence of hemolysis or hepatic pathology), who will be allowed only in consultation with their physician, AND ALT (SGPT) and/or AST (SGOT) ≤2.5 x ULN

Exclusion criteria:

* Pathogenic POLE mutation(s)
* Mismatch repair deficiency
* Major surgical procedure (as defined by the investigator) within 28 days prior to the first dose of the IP
* History of allogenic organ transplantation
* Uncontrolled intercurrent illness, including but not limited to, ongoing or active infection, symptomatic congestive heart failure, uncontrolled hypertension, unstable angina pectoris, cardiac arrhythmia, interstitial lung disease, serious chronic gastrointestinal conditions associated with diarrhea, or psychiatric illness/social situations that would limit compliance with study requirement, substantially increase risk of incurring AEs or compromise the ability of the patient to give written informed consent
* Any previous treatment with a PARP inhibitor, including olaparib
* History of active primary immunodeficiency
* History or evidence of hemorrhagic disorders within 6 months prior to randomization
* Patients with myelodysplastic syndrome/acute myeloid leukemia history or with features suggestive of MDS/AML
* Previous allogenic bone marrow transplant or double umbilical cord blood transplantation (dUCBT)
* Active infection, including: tuberculosis (clinical evaluation that includes clinical history, physical examination and radiographic findings, and TB testing in line with local practice), hepatitis B (known positive HBV surface antigen (HBsAg) result), hepatitis C, or human immuno-deficiency virus (positive HIV 1/2 antibodies). Patients with a past or resolved HBV infection (defined as the presence of hepatitis B core antibody [anti-HBc] and absence of HBsAg) are eligible. Patients positive for hepatitis C (HCV) antibody are eligible only if polymerase chain reaction is negative for HCV RNA.
* Concomitant use of known strong CYP3A inhibitors (eg. itraconazole, telithromycin, clarithromycin, protease inhibitors boosted with ritonavir or cobicistat, indinavir, saquinavir, nelfinavir, boceprevir, telaprevir) or moderate CYP3A inhibitors (eg. ciprofloxacin, erythromycin, diltiazem, fluconazole, verapamil). The required washout period prior to starting olaparib is 2 weeks.
* Concomitant use of known strong (eg. phenobarbital, enzalutamide, phenytoin, rifampicin, rifabutin, rifapentine, carbamazepine, nevirapine and St John's Wort) or moderate CYP3A inducers (eg. bosentan, efavirenz, modafinil). The required washout period prior to starting olaparib is 5 weeks for enzalutamide or phenobarbital and 3 weeks for other agents.
* Patients unable to swallow orally administered medication and patients with gastrointestinal disorders likely to interfere with absorption of the study medication.
* Medical or psychological condition which in the opinion of the investigator would not permit the patient to complete the study or sign meaningful informed consent.

The MMRd-GREEN trial

Inclusion criteria:

* Mismatch repair deficient EC
* Histologically confirmed (FIGO 2009) stage IB/II EC with myometrial or cervical stroma involvement and lympovascular space invasion (LVSI) OR Stage III EC OR Stage IVA with limited pelvic peritoneal involvement
* WHO Performance score 0-1
* Body weight > 30 kg
* Adequate systemic organ function:

  * Creatinine clearance (> 40 cc/min): Measured creatinine clearance (CL) >40 mL/min or Calculated creatinine CL>40 mL/min by the Cockcroft-Gault formula (Cockcroft and Gault 1976) or by 24-hour urine collection for determination of creatinine clearance.
  * Adequate bone marrow function : hemoglobin >9.0 g/dl, Absolute neutrophil count (ANC) ≥1.0 x 109/l, platelet count ≥75 x 109/l.
  * Adequate liver function: bilirubin ≤1.5 x institutional upper limit of normal (ULN). <<This will not apply to patients with confirmed Gilbert's syndrome (persistent or recurrent hyperbilirubinemia that is predominantly unconjugated in the absence of hemolysis or hepatic pathology), who will be allowed only in consultation with their physician.>> AND ALT (SGPT) and/or AST (SGOT) ≤2.5 x ULN

Exclusion criteria:

* Pathogenic POLE mutation(s)
* Major surgical procedure (as defined by the Investigator) within 28 days prior to the first dose of investigational medicinal product (IMP)
* History of allogenic organ transplantation
* Uncontrolled intercurrent illness, including but not limited to, ongoing or active infection, symptomatic congestive heart failure, uncontrolled hypertension, unstable angina pectoris, cardiac arrhythmia, interstitial lung disease, serious chronic gastrointestinal conditions associated with diarrhea, or psychiatric illness/social situations that would limit compliance with study requirement, substantially increase risk of incurring AEs or compromise the ability of the patient to give written informed consent.
* Any previous treatment with a PD(L)1 inhibitor, including durvalumab.
* Receipt of live attenuated vaccine within 30 days prior to the first dose of durvalumab. Note: Patients, if enrolled, should not receive live vaccine whilst receiving IP and up to 30 days after the last dose of IMP.
* Current or prior use of immunosuppressive medication within 14 days before the first dose of durvalumab with the exceptions of:

  * Intranasal, inhaled, topical steroids, or local steroid injections (e.g., intra articular injection).
  * Systemic corticosteroids at physiologic doses not to exceed <<10 mg/day>> of prednisone or its equivalent.
  * Steroids as premedication for hypersensitivity reactions (e.g., CT scan premedication).
* History of active primary immunodeficiency
* Active or prior documented autoimmune or inflammatory disorders (including inflammatory bowel disease [e.g., colitis or Crohn's disease], diverticulitis [with the exception of diverticulosis], systemic lupus erythematosus, Sarcoidosis syndrome, or Wegener syndrome. The following are exceptions to this criterion:

  * Patients with vitiligo or alopecia
  * Patients with hypothyroidism (e.g., following Hashimoto syndrome)stable on hormone replacement
  * Any chronic skin condition that does not require systemic therapy
  * Patients without active disease in the last 5 years may be included but only after consultation with the study physician.
* Active infection including tuberculosis (clinical evaluation that includes clinical history, physical examination and radiographic findings, and TB testing in line with local practice), hepatitis B (known positive HBV surface antigen (HBsAg) result), hepatitis C, or human immuno-deficiency virus (positive HIV 1/2 antibodies). Patients with a past or resolved HBV infection (defined as the presence of hepatitis B core antibody [anti-HBc] and absence of HBsAg) are eligible. Patients positive for hepatitis C (HCV) antibody are eligible only if polymerase chain reaction is negative for HCV RNA.
* Medical or psychological condition which in the opinion of the investigator would not permit the patient to complete the study or sign meaningful informed consent.

The NSMP-ORANGE trial

Inclusion criteria:

* NSMP EC
* Histologically confirmed stage II EC with substantial LVSI or stage III EC
* ER positive EC
* WHO performance status 0-1

Exclusion criteria:

* Pathogenic POLE mutation(s)
* Mismatch repair deficiency
* p53 abnormality

The POLEmut-BLUE trial

Inclusion criteria:

* Pathogenic POLE mutation(s)
* For the main cohort, patients must have one of the following combinations of FIGO stage, grade, and LVSI:

  * stage IA (not confined to polyp), grade 3, pN0, with or without LVSI
  * stage IB, grade 1 or 2, pNx/N0, with or without LVSI
  * stage IB, grade 3, pN0, without substantial LVSI
  * stage II (microscopic), grade 1 or 2, pN0, without substantial LVSI
* For the exploratory cohort, patients must have one of the following combinations of FIGO stage, grade, and LVSI:

  * stage IA (not confined to polyp), grade 3 - Stage III not included in main cohort
  * Multiple molecular classifiers stage IA (not confined to polyp), grade 3 - Stage III
* Patient consent must be appropriately obtained in accordance with applicable local and regulatory requirements. Each patient must sign a consent form prior to enrolment in the trial to document their willingness to participate. A similar process must be followed for sites outside of Canada as per their respective cooperative group's procedures.
* Patient is able (i.e., sufficiently fluent) and willing to complete the QOL and/or health utility questionnaires in either English, French or a validated language. The baseline assessment must be completed within the required timelines, prior to enrolment. Inability (lack of comprehension in English or French, or other equivalent reason such as cognitive issues or lack of competency) to complete the questionnaires will not make the patient ineligible for the study. However, ability but unwillingness to complete the questionnaires will make the patient ineligible.
* Patients must be accessible for treatment and follow up. Patients enrolled on this trial must be treated and followed at the participating center. Investigators must assure themselves the patients enrolled on this trial will be available for complete documentation of the treatment, adverse events, and follow-up.
* Patients must agree to return to their primary care facility for any adverse events which may occur through the course of the trial.
* In accordance with CCTG policy, protocol treatment is to begin within 10 weeks of hysterectomy/bilateral salpingo-oophorectomy.

Exclusion criteria:

* Prior chemotherapy for EC
* Isolated tumor cells identified in lymph node(s) for main study cohort (patient can be included in exploratory cohort)

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes — Female sex
Enrollment: 1615 (Estimated)
Dates: Start 2021-11-11 (Actual); Primary Completion 2030-01-01 (Estimated); Study Completion 2031-01-01 (Estimated)

PRIMARY OUTCOMES:
p53abn-RED trial | 3 years
  Recurrence-free survival
MMRd-GREEN trial | 3 years
  Recurrence-free survival
NSMP-ORANGE trial | 3 years
  Recurrence-free survival
POLEmut-BLUE trial | 3 years
  Pelvic recurrence-free survival

SECONDARY OUTCOMES:
Recurrence-free survival | 5 years
  All RAINBO trials
Pelvic recurrence-free survival | 5 years
  All RAINBO trials
Vaginal recurrence-free survival | 3 years, 5 years
  All RAINBO trials
Endometrial cancer-specific survival | 3 years, 5 years
  All RAINBO trials
Overall survival | 3 years, 5 years
  All RAINBO trials
Treatment-related toxicity - according to CTCAE v5.0 | 3 years, 5 years
  All RAINBO trials
Health-related quality of life - Assessed using the EORTC QLQ-C30 questionnaire | 3 years, 5 years
  All RAINBO trials
Health-related quality of life - Assessed using the EORTC QLQ-EN24 questionnaire | 3 years, 5 years
  All RAINBO trials

CONTACTS AND LOCATIONS:
Overall Officials: Alexandra Leary, Md PhD, Principal Investigator — Institute Gustave Roussy, Villejuif, France (p53abn-RED trial); Judith R Kroep, MD PhD, Principal Investigator — Leiden University Medical Center, Leiden, The Netherlands (MMRd-GREEN trial); Melanie E Powell, Md PhD, Principal Investigator — Barts Health NHS Trust, London, United Kingdom (NSMP-ORANGE trial); Emma J Crosbie, Md PhD, Principal Investigator — St Mary's Hospital, Manchester, United Kingdom (NSMP-ORANGE trial); Kathy Han, Md PhD, Principal Investigator — Princess Margaret Cancer Centre, University of Toronto, Toronto, Canada (POLEmut-BLUE trial); Jessica N McAlpine, Md PhD, Principal Investigator — University of British Columbia,Vancouver, Canada (POLEmut-BLUE trial)
Locations (14):
- Canada (2):
  - The POLEmut-BLUE trial: Princess Margaret Cancer Centre, University of Toronto, Toronto
  - The POLEmut-BLUE trial: University of British Columbia, Vancouver
- The p53abn-RED trial: Institute Gustave Roussy, Villejuif, France
- Netherlands (9):
  - Amsterdam University Medical Center, Amsterdam
  - Amphia Ziekenhuis, Breda
  - Instituut Verbeeten, Breda
  - Catharina Ziekenhuis, Eindhoven
  - Medisch Spectrum Twente, Enschede
  - Universitair Medisch Centrum Groningen, Groningen
  - The MMRd-GREEN trial: Leiden University Medical Center, Leiden
  - Erasmus Medical Center, Rotterdam
  - Haags Medisch Centrum, The Hague
- United Kingdom (2):
  - The NSMP-ORANGE trial: Barts Health NHS Trust, London
  - The NSMP-ORANGE trial: Manchester Academic Health Science Centre, St Mary's Hospita, Manchester

IPD SHARING:
Plan to Share IPD: Yes
Following the planned translational work in the RAINBO programme and publications, the translational research (TR) committee will open up the sample collection to external researchers. Access will be granted following completion of a research proposal form and approval by the TR committee chaired by Dr. Tjalling Bosse. All external researchers will be expected to demonstrate funding for their project and ethics approval. Data will be made available as required through data sharing agreements. The following will be reviewed when considering applications for data sharing and sample access: data and sample use is in-keeping with patient consent, the proposed project has scientific value, with defined objectives and study plan, trial data are appropriate for the intended purpose, acknowledgement of the RAINBO Programme in all publications that arise from the data sharing, compliance with legal and regulatory requirements as applicable and patient confidentiality maintained at all times.
Supporting Information: Study Protocol
Time Frame: The study protocols of the four trials will be made made available on the trial's websites by the time the trials open
Access Criteria: Public

REFERENCES:
- [Background] IMPLEMENTATION OF COLLABORATIVE TRANSLATIONAL RESEARCH (TRANSPORTEC) FINDINGS IN AN INTERNATIONAL ENDOMETRIAL CANCER CLINICAL TRIALS PROGRAM (RAINBO). T Bosse, M Powell, E Crosbie, A Leary, J Kroep, K Han, J Mcalpine, N Horeweg, S De Boer, M De Bruyn, R Nout, V Smit, HW Nijman, N Singh, H Mackay, R Edmondson, L Mileshkin, D Church, H Kitchener, CL Creutzberg. Int J Gynecol Cancer 2021;31(Suppl 3):A1-A395. DOI: 10.1136/ijgc-2021-ESGO.171
- [Background] RAINBO Research Consortium. Refining adjuvant treatment in endometrial cancer based on molecular features: the RAINBO clinical trial program. Int J Gynecol Cancer. 2023 Jan 3;33(1):109-117. doi: 10.1136/ijgc-2022-004039. PMID 36600534
- [Derived] Secord AA, Powell MA, McAlpine J. Molecular Characterization and Clinical Implications of Endometrial Cancer. Obstet Gynecol. 2025 Nov 1;146(5):660-671. doi: 10.1097/AOG.0000000000006080. Epub 2025 Sep 18. PMID 40966692